CLINICAL TRIAL: NCT02270983
Title: A Phase 2 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Trial of Linaclotide Administered Orally for 8 Weeks to Adult Outpatients With Opioid-Induced Constipation Receiving Chronic Opioid Treatment for Non-Cancer Pain
Brief Title: Phase 2 Randomized, Double-Blind, Placebo-Controlled, Parallel Group Trial of Linaclotide Administered to Patients With Opioid-Induced Constipation Receiving Chronic Opioid Treatment for Non-Cancer Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIN-MD-40
Record Dates: First submitted 2014-10-16; First posted 2014-10-22 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Opioid-Induced Constipation
Keywords: Opioid-Induced Constipation; Linaclotide; Linzess
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Linaclotide 145 micrograms (Experimental): Oral capsule, taken once daily each morning at least 30 minutes before breakfast, with the exception of the first Treatment Period dose which will be taken at the study center after at least a 2-hour fast.
  Interventions: Drug: Linaclotide 145 micrograms
- Linaclotide 290 micrograms (Experimental): Oral capsule, taken once daily each morning at least 30 minutes before breakfast, with the exception of the first Treatment Period dose which will be taken at the study center after at least a 2-hour fast.
  Interventions: Drug: Linaclotide 290 micrograms
- Placebo (Experimental): Oral capsule, taken once daily each morning at least 30 minutes before breakfast, with the exception of the first Treatment Period dose which will be taken at the study center after at least a 2-hour fast.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linaclotide 145 micrograms
  Other Names: Linzess
  Arms: Linaclotide 145 micrograms
Drug: Linaclotide 290 micrograms
  Other Names: Linzess
  Arms: Linaclotide 290 micrograms
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of linaclotide for the treatment of opioid-induced constipation (OIC), in adults receiving stable opioid treatment for chronic non-cancer pain that has been present for a minimum of 3 months.

This study included up to a 4-week Screening Period, and a 2 to 3-week Pretreatment Period. Patients meeting the entry criteria were randomized to 1 of 2 doses of linaclotide or placebo once per day for 8 weeks. This 8-week study assessed the effects of linaclotide on bowel movement frequency, as well as other bowel symptoms of OIC.

ELIGIBILITY:
Inclusion Criteria:

* Patient has chronic non-cancer pain that has been present for a minimum of 3 months
* Patient has been receiving a stable oral dose of a full-opioid agonist for at least 4 days per week during the 8 consecutive weeks
* Patient meets protocol criteria for Opioid-Induced Constipation (OIC): < 3 spontaneous bowel movements (SBMs) per week and reports one of the following symptoms for at least 4 weeks:

  1. Straining during > 25% of BMs
  2. Lumpy or hard stools during > 25% of BMs
  3. Sensation of incomplete evacuation during > 25% of BMs
* Patient meets the colonoscopy requirements defined by the American Gastroenterological Association guidelines
* Patient has successfully completed protocol procedures (with no clinically significant findings)
* Patient is compliant with Interactive Voice Response System (IVRS) for daily diary reporting
* Patient has a total of < 6 SBMs in IVRS during the 14 days before and up to the time of Randomization
* Patient has adequate relief and well-controlled pain with current dose of opioid

Exclusion Criteria:

* Patient has been using opioids for abdominal pain
* Patient has symptoms of or been diagnosed with chronic constipation or chronic idiopathic constipation prior to initiation of opioid treatment
* Patient has symptoms of or been diagnosed with Irritable Bowel Syndrome (IBS) prior to initiation of opioid treatment
* Patient has a history of loose or watery stools for > 25% of BMs during the 3 months before the Screening in the absence of laxatives, suppositories, or enemas
* Patient has a structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility
* Patient has any protocol-excluded or clinically significant medical or surgical history that would limit the patient's ability to complete or participate in this clinical trial or could confound the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia D'Astoli, RN, Study Director — Forest Laboratories, LLC, an Allergan Affiliate
Locations (77):
- United States (77):
  - Forest Investigative Site 002, Anniston, Alabama
  - Forest Investigative Site 001, Foley, Alabama
  - Forest Investigative Site 007, Phoenix, Arizona
  - Forest Investigative Site 008, Tucson, Arizona
  - Forest Investigative Site 003, North Little Rock, Arkansas
  - Forest Investigative Site 018, Anaheim, California
  - Forest Investigative Site 014, Fountain Valley, California
  - Forest Investigative Site 019, Fresno, California
  - Forest Investigative Site 017, Garden Grove, California
  - Forest Investigative Site 010, Gold River, California
  - Forest Investigative Site 009, Lincoln, California
  - Forest Investigative Site 012, North Hollywood, California
  - Forest Investigative Site 011, Orange, California
  - Forest Investigative Site 016, Sacramento, California
  - Forest Investigative Site 013, San Diego, California
  - Forest Investigative Site 015, Santa Ana, California
  - Forest Investigative Site 020, Colorado Springs, Colorado
  - Forest Investigative Site 021, Bristol, Connecticut
  - Forest Investigative Site 035, Boynton Beach, Florida
  - Forest Investigative Site 038, Bradenton, Florida
  - Forest Investigative Site 024, DeLand, Florida
  - Forest Investigative Site 027, Gainesville, Florida
  - Forest Investigative Site 023, Jacksonville, Florida
  - Forest Investigative Site 036, Jupiter, Florida
  - Forest Investigative Site 037, Lauderdale Lakes, Florida
  - Forest Investigative Site 028, Miami, Florida
  - Forest Investigative Site 040, Orlando, Florida
  - Forest Investigative Site 022, Oviedo, Florida
  - Forest Investigative Site 034, Port Orange, Florida
  - Forest Investigative Site 029, Seminole, Florida
  - Forest Investigative Site 031, Tampa, Florida
  - Forest Investigative Site 033, Tampa, Florida
  - Forest Investigative Site 030, Tampa, Florida
  - Forest Investigative Site 039, West Palm Beach, Florida
  - Forest Investigative Site 032, Weston, Florida
  - Forest Investigative Site 041, Marietta, Georgia
  - Forest Investigative Site 042, Woodstock, Georgia
  - Forest Investigative Site 043, Chicago, Illinois
  - Forest Investigative Site 044, Evansville, Indiana
  - Forest Investigative Site 045, Madisonville, Kentucky
  - Forest Investigative Site 046, Metairie, Louisiana
  - Forest Investigative Site 048, Hagerstown, Maryland
  - Forest Investigative Site 047, Watertown, Massachusetts
  - Forest Investigative Site 050, Chesterfield, Michigan
  - Forest Investigative Site 049, Flint, Michigan
  - Forest Investigative Site 058, Omaha, Nebraska
  - Forest Investigative Site 057, Omaha, Nebraska
  - Forest Investigative Site 059, Williamsville, New York
  - Forest Investigative Site 082, Asheboro, North Carolina
  - Forest Investigative Site 054, Chapel Hill, North Carolina
  - Forest Investigative Site 088, Davidson, North Carolina
  - Forest Investigative Site 051, Flat Rock, North Carolina
  - Forest Investigative Site 052, Greensboro, North Carolina
  - Forest Investigative Site 055, Greensboro, North Carolina
  - Forest Investigative Site 053, Winston-Salem, North Carolina
  - Forest Investigative Site 056, Fargo, North Dakota
  - Forest Investigative Site 062, Cincinnati, Ohio
  - Forest Investigative Site 061, Columbus, Ohio
  - Forest Investigative Site 060, Mentor, Ohio
  - Forest Investigative Site 087, Wadsworth, Ohio
  - Forest Investigative Site 064, Oklahoma City, Oklahoma
  - Forest Investigative Site 063, Oklahoma City, Oklahoma
  - Forest Investigative Site 065, Tulsa, Oklahoma
  - Forest Investigative Site 066, Medford, Oregon
  - Forest Investigative Site 067, Levittown, Pennsylvania
  - Forest Investigative Site 080, Philadelphia, Pennsylvania
  - Forest Investigative Site 068, Cumberland, Rhode Island
  - Forest Investigative Site 070, Charleston, South Carolina
  - Forest Investigative Site 083, Richardson, Texas
  - Forest Investigative Site 074, San Antonio, Texas
  - Forest Investigative Site 073, San Antonio, Texas
  - Forest Investigative Site 071, San Antonio, Texas
  - Forest Investigative Site 075, Logan, Utah
  - Forest Investigative Site 084, Ogden, Utah
  - Forest Investigative Site 076, West Jordan, Utah
  - Forest Investigative Site 078, Christiansburg, Virginia
  - Forest Investigative Site 079, Bellevue, Washington

REFERENCES:
- [Derived] Brenner DM, Argoff CE, Fox SM, Bochenek W, D'Astoli P, Blakesley RE, Reasner DS, O'Dea CR, Cash BD. Efficacy and safety of linaclotide for opioid-induced constipation in patients with chronic noncancer pain syndromes from a phase 2 randomized study. Pain. 2020 May;161(5):1027-1036. doi: 10.1097/j.pain.0000000000001754. PMID 32310620

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 calendar days (minimum) to 21 calendar days (maximum) before randomization, participants had to provide information about bowel habits, symptom severity, and rescue medication use through daily IVRS calls. A total of 254 patients were randomized to treatment.
Period: Overall Study
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Started | 79 | 87 | 88
Completed | 70 | 80 | 76
Not Completed | 9 | 7 | 12
Not completed — Adverse Event | 3 | 2 | 6
Not completed — Lack of Efficacy | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — family emergency | 0 | 1 | 0
Not completed — study procedure non-compliance | 1 | 0 | 0
Not completed — moved away from study site | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Of the 254 participants who were randomized to treatment, 2 patients were randomized in error and did not receive investigational product. 252 of the randomized participants did receive investigational product and comprise the Safety and ITT populations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms | Total
Number analyzed (Participants) | 78 | 87 | 87 | 252
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (10.6) | 53.1 (9.2) | 54.0 (10.5) | 53.2 (10.1)
Age, Customized [Count of Participants; unit: Participants]
  18 to under 40 | 11 | 4 | 6 | 21
  40 to under 65 | 56 | 71 | 67 | 194
  65 and over | 11 | 12 | 14 | 37
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 31 | 38 | 32 | 101
  Female | 47 | 49 | 55 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 66 | 71 | 72 | 209
  Race: Black or African American | 9 | 15 | 10 | 34
  Race: Asian | 3 | 1 | 3 | 7
  Race: American Indian or Alaska Native | 0 | 0 | 1 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Multiple Races | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 4 | 5 | 2 | 11
  Ethnicity: Not Hispanic or Latino | 74 | 82 | 85 | 241
Weight [Mean (Standard Deviation); unit: kg] | 90.64 (24.56) | 85.45 (22.78) | 89.78 (22.61) | 88.55 (23.31)
Height [Mean (Standard Deviation); unit: cm] | 168.05 (12.27) | 170.70 (10.17) | 168.00 (10.62) | 168.95 (11.04)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.17 (8.57) | 29.09 (6.32) | 31.77 (7.39) | 30.97 (7.54)
SBM Frequency Rate [Mean (Standard Deviation); unit: SBMs per week] — Number of spontaneous bowel movements (SBMs) per week
  SBMs per week | 1.05 (0.81) | 1.01 (0.70) | 1.14 (0.84) | 1.07 (0.78)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 8-Week SBM Frequency Rate (SBMs/Week)
Description: Change from baseline in 8-Week SBM frequency rate (SBMs/week) during the Treatment Period.
Time Frame: Baseline (Week 0) to Week 8
Population: 252 participants received at least one dose of study drug, comprising the ITT study population.
Measure: Least Squares Mean (Standard Error); unit: Number of SBMs per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 78 | 87 | 87
Number of SBMs per week | 1.474 (0.361) | 2.799 (0.350) | 3.382 (0.353)
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 145 Micrograms; Test type: Superiority; p = 0.0035, ANCOVA; Least squares mean difference = 1.325, 95% CI 2-sided [0.439 to 2.211], Standard Error of Mean 0.450
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290 Micrograms; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = 1.908, 95% CI 2-sided [1.021 to 2.796], Standard Error of Mean 0.451

2. Secondary Outcome: Time to First SBM After the First Dose of Investigational Product
Description: The median time to the first SBM after the first dose of investigational product
Time Frame: Baseline (Day 0) up to 8 weeks
Population: 252 participants received at least one dose of study drug, comprising the ITT study population.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 78 | 87 | 87
hours | 47.1 [25.0 to 71.8] | 26.5 [21.8 to 45.0] | 28.7 [23.5 to 47.0]
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 145 Micrograms; Test type: Superiority; p = 0.1429, Log Rank; Cox Proportional Hazard = 1.28, 95% CI 2-sided [0.92 to 1.77]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290 Micrograms; Test type: Superiority; p = 0.0287, Log Rank; Cox Proportional Hazard = 1.43, 95% CI 2-sided [1.04 to 1.97]

3. Secondary Outcome: Percentage of Participants Meeting 6/8 Week Spontaneous Bowel Movement (SBM) 3 + 1 Responder Criteria
Description: A 6/8 Week SBM 3 + 1 responder was a participant who met the weekly SBM 3 + 1 responder criteria for at least 6 out of the 8 weeks of the Treatment Period. For each week in the Treatment Period, a weekly SBM 3 + 1 responder was a patient who had an SBM weekly rate ≥ 3 and an increase ≥ 1 in the SBM weekly rate from baseline for that week.
Time Frame: 8-week treatment period
Population: 252 participants received at least one dose of study drug, comprising the ITT study population.
Measure: Number; unit: Percentage of Responders
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 78 | 87 | 87
Percentage of Responders | 33.3 | 40.2 | 47.1
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 145 Micrograms; Test type: Superiority; p = 0.3332, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel tests comparing specified treatment groups, controlling for geographic region; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.73 to 2.58]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290 Micrograms; Test type: Superiority; p = 0.0506, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel tests comparing specified treatment groups, controlling for geographic region; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.00 to 3.68]

4. Secondary Outcome: Change From Baseline in 8-Week Stool Consistency
Description: Stool Consistency was assessed using the 7-Point Bristol Stool Form Scale:
  1. = separate hard lumps like nuts (difficult to pass)
  2. = sausage shaped but lumpy
  3. = like a sausage but with cracks on surface
  4. = like a sausage or snake, smooth and soft
  5. = soft blobs with clear-cut edges (passed easily)
  6. = fluffy pieces with ragged edges, a mushy
  7. = watery, no solid pieces (entirely liquid)
Time Frame: Baseline (Week 0) to Week 8
Population: Of the 252 participants in the ITT population, 200 participants had Stool Consistency data collected
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 59 | 71 | 70
Units on a scale | 0.911 (0.172) | 1.662 (0.165) | 1.898 (0.168)
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 145 Micrograms; Test type: Superiority; p = 0.0007, ANCOVA; Least squares mean difference = 0.751, 95% CI 2-sided [0.324 to 1.178], Standard Error of Mean 0.217
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290 Micrograms; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = 0.987, 95% CI 2-sided [0.558 to 1.416], Standard Error of Mean 0.217

5. Secondary Outcome: Change From Baseline in 8-Week Straining
Description: Straining was measured on a 5-point ordinal scale where a value of 1 is "not at all" and a value of 5 is "an extreme amount."
Time Frame: Baseline (Week 0) to Week 8
Population: Of the 252 participants in the ITT population, 200 participants had 8-week straining data collected
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 59 | 71 | 70
Units on a scale | -0.753 (0.116) | -1.212 (0.111) | -1.422 (0.112)
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 145 Micrograms; Test type: Superiority; p = 0.0017, ANCOVA; Least squares mean difference = -0.460, 95% CI 2-sided [-0.746 to -0.174], Standard Error of Mean 0.145
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290 Micrograms; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -0.669, 95% CI 2-sided [-0.957 to -0.382], Standard Error of Mean 0.146

6. Secondary Outcome: Change From Baseline in 8-Week Abdominal Bloating
Description: Abdominal bloating was collected daily via IVRS calls and measured using an 11-point numerical rating scale, where 0 represents no abdominal bloating and 10 represents very severe abdominal bloating.
Time Frame: Baseline (Week 0) to Week 8
Population: 252 participants received at least one dose of study drug, comprising the ITT study population.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 78 | 87 | 87
Units on a scale | -0.983 (0.164) | -0.950 (0.160) | -1.590 (0.160)
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 145 Micrograms; Test type: Superiority; p = 0.8720, ANCOVA; Least squares mean difference = 0.033, 95% CI 2-sided [-0.371 to 0.437], Standard Error of Mean 0.205
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290 Micrograms; Test type: Superiority; p = 0.0034, ANCOVA; Least squares mean difference = -0.607, 95% CI 2-sided [-1.011 to -0.203], Standard Error of Mean 0.205

ADVERSE EVENTS:
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
All-Cause Mortality (participants affected / at risk) | 1/78 | 0/87 | 0/87
Serious Adverse Events (participants affected / at risk) | 5/78 | 0/87 | 1/87
Other Adverse Events (participants affected / at risk) | 16/78 | 24/87 | 33/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=78) | Linaclotide 145 Micrograms (N=87) | Linaclotide 290 Micrograms (N=87)
Seizure (Nervous system disorders) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transient Ischaemic Attack (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=78) | Linaclotide 145 Micrograms (N=87) | Linaclotide 290 Micrograms (N=87)
Diarrhoea (Gastrointestinal disorders) | 13 | 24 | 32
Nausea (Gastrointestinal disorders) | 4 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the Investigator will be subject to mutual agreement between the Investigator, Forest Research Institute, Inc., an affiliate of Allergan, and Ironwood Pharmaceuticals Inc.